CLINICAL TRIAL: NCT05300607
Title: The Western Ontario Rotator Cuff Index Arabic Version: Cross-cultural Adaptation, Validity, and Reliability for Patients With Rotator Cuff Disease
Brief Title: The Western Ontario Rotator Cuff Index Arabic Version
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Lydia Nasser Zaki, Principal Investigator, Cairo University
Other Study IDs: P.T.REC/012/003550
Record Dates: First submitted 2022-02-05; First posted 2022-03-29 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Surveys and Questionnaires; Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- questionnaire: rotator cuff diseases patients will self report the items of the Arabic version of The Western Ontario Rotator Cuff Index questionnaire
  Interventions: Other: Cross-cultural adaptation, validity, and reliability

INTERVENTIONS:
Other: Cross-cultural adaptation, validity, and reliability — evaluation, translation, cultural adaption, validation, and investigation of the reliability of Arabic version of The Western Ontario Rotator Cuff Index (WORC) to be used in Arabic countries.

SUMMARY:
To evaluate, translate, culturally adapt, validate, and investigate the reliability of Arabic version of The Western Ontario Rotator Cuff Index (WORC).

The null hypothesis of this study will be stated as:

Arabic language version of the WORC doesn't have face, content, or construct validity enough to measure quality of life related to rotator cuff disorders in Arabic patients.

Arabic language version of the WORC doesn't have reliability to measure quality of life related to rotator cuff disorders in Arabic patients

DETAILED DESCRIPTION:
The WORC is an increasingly applied outcome measure for rotator cuff conditions. The WORC is a self-assessment scale that was developed to measure the quality of life of patients with RC disorders. It contains 21 items representing 5 subscales: physical symptoms 6 items, sports/recreation 4 items, work 4 items, lifestyle 4 items, and emotions 3 items, which encompass all aspects of heath as defined by the World Health Organization.

It has been translated and validated in several languages, including Chinese, Dutch, French-Canadian, Japanese, Norwegian, Persian, Polish, Portuguese - Brazilian, Spanish, Swedish and Turkish.

The current studies point out the increasing need for a questionnaire specifically developed to measure health related quality of life in patients treated conservatively, and respecting the following main characteristics: presenting adequate measurement properties and allowing to make comparisons of health-related quality of life between patients.

Cross-cultural adaptation allows globalization of information worldwide without the loss of the conceptual meaning. This enables the exchange and comparisons of valid information among different populations worldwide.

The Western Ontario Rotator Cuff Index has not been translated into the Arabic language, so it has a limited use in Egypt as well as Arabic countries. Therefore, the aim of this study is to translate, culturally adapt, validate, and investigate the reliability of Arabic version of The Western Ontario Rotator Cuff Index.

ELIGIBILITY:
Inclusion Criteria:

* Referred with rotator cuff tendinopathy or rotator cuff partial tear by physician.
* Able to read and write in Arabic.
* Their age will be Between 18 to 60 years old
* patients with chronic inflammatory diseases will be included

Exclusion Criteria:

* Patients with impairments in the cervical spine, elbow, or hand affecting the shoulder function
* Patients that have Cognitive alterations
* Patients that have any systemic disease that may affect patient's outcome.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with rotator cuff diseases from outpatient clinics
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
Translation of western Ontario rotator cuff index questionnaire into Arabic for patients with rotator cuff injuries | 6 months
  It will be performed according to the guidelines of Sousa. First forward translation of the questionnaire from English to Arabic producing two forward-translated versions of the questionnaire then the instructions, the items and the response format of the forward-translated versions are compared for any discrepancies that must be discussed and resolved using expert committee. then the translated Arabic version will be Back-translated to English producing two back-translated versions. then the instructions, items, and response format of both the two back-translations and the original questionnaire are compared by expert committee regarding format, grammatical structure, similarity in meaning, and relevance to derive a pre-final version of the questionnaire in Arabic. This version is pilot tested among participants whose language is Arabic to evaluate questionnaire for clarity. Participants should be recruited from the target population of the questionnaire
Validation of Arabic version of The Western Ontario Rotator Cuff Index questionnaire for patients with rotator cuff injuries | 6 months
  The Disabilities of the Arm, Shoulder and Hand questionnaire and The Short Form 36 questionnaire will be used for the validity process to establish correlation between the subscales of Western Ontario Rotator Cuff Index questionnaire and the subscales of The Disabilities of the Arm, Shoulder and Hand questionnaire and The Short Form 36 questionnaire which has already been translated and validated in its Arabic version.
  Concurrent validity will be evaluated by comparing Western Ontario Rotator Cuff Index questionnaire domains with relevant domains in The Disabilities of the Arm, Shoulder and Hand questionnaire and The Short Form 36 questionnaire The western Ontario rotator cuff index questionnaire consists of 21 items Each item is answered on a 100 - mm visual analog scale. 0 is minimum score and 100 is maximum score. The scores of 21 items are added to give a total score from 0 to 2100.The highest or most symptomatic score is 2100, and the best or asymptomatic score is 0
Establishing the full psychometric properties of the Arabic version of the western Ontario rotator cuff index questionnaire for patients with rotator cuff injuries | 6 months
  The questionnaire has 21 items with 5 domains: physical symptoms(6 items), sport(4 items), work(4 items), lifestyle(4 items), and emotional(3 items). It has instructions to the patients and a supplement with an explanation of each item. Each item is answered on a 100 - mm visual analog scale, 0 is minimum and 100 is maximum score. The scores of 21 items are added to give a total from 0 to 2100.The highest or most symptomatic score is 2100, and the best or asymptomatic score is 0. 200 patients with rotator cuff injuries will participate. Patients will fill out the Arabic version of western Ontario rotator cuff index questionnaire along with the Arabic version of both the Short Form 36 questionnaire and Disabilities, of the Arm, Shoulder, and Hand questionnaire and 1 week later, the patient will refill out the 3 questionnaires. the short form 36, Disabilities, of the Arm, Shoulder, and Hand and the western Ontario rotator cuff index questionnaires contain similar subscales.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser M. Aneis, PHD, Study Director — Cairo University; Mohsen El Sayyad, PHD, Study Chair — Cairo University
Locations (1):
- Faculty of physical therapy basic science department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing the results and the Arabic version of the questionnaire to be available to be used with rotator cuff diseases patients in Arabic countries
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: the Arabic version will be shared with Arabic countries medical stuff who tend to measure the quality of life of patients with rotator cuff diseases

REFERENCES:
- [Background] Kirkley A, Alvarez C, Griffin S. The development and evaluation of a disease-specific quality-of-life questionnaire for disorders of the rotator cuff: The Western Ontario Rotator Cuff Index. Clin J Sport Med. 2003 Mar;13(2):84-92. doi: 10.1097/00042752-200303000-00004. PMID 12629425
- [Background] Sousa VD, Rojjanasrirat W. Translation, adaptation and validation of instruments or scales for use in cross-cultural health care research: a clear and user-friendly guideline. J Eval Clin Pract. 2011 Apr;17(2):268-74. doi: 10.1111/j.1365-2753.2010.01434.x. Epub 2010 Sep 28. PMID 20874835